CLINICAL TRIAL: NCT01268813
Title: Personalized Medicine in Diabetes Using a Nanotechnology Platform
Brief Title: Personalized Medicine for Diabetes Prediction and Prevention of Complications
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Prof. Eddy Karnieli, Rambam Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: METASC011
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-11

CONDITIONS: Metabolic Syndrome; Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exhaled breath uptake blood test (Experimental): Diabetic patients receiving oral hypoglycemic drug will be tested for biomarkers in their breath and blood samples
  Interventions: Other: Breath analysis and blood analysis
- Exhaled breath and blood test (No Intervention): Breath and blood samples will be collected from healthy volunteers and analyzed using Gas Chromatography-Mass Spectroscopy. The results will be compared to the experimental arm.
  Interventions: Other: Breath analysis and blood analysis

INTERVENTIONS:
Other: Breath analysis and blood analysis — Exhaled breath and blood samples will be collected and further tested using Gas Chromatography-Mass Spectroscopy system.
  Other Names: nanothecnology platform

SUMMARY:
The metabolic syndrome is a collection of related risk factors that predispose to the development of type 2 diabetes Mellitus and cardiovascular disease. The investigators will examine the hypothesis that the metabolic and genomic characteristics of patients with metabolic syndrome and/or diabetes that are at risk for developing complications differ from each other and can be detected using specific biomarkers in blood or in the exhaled breath. Early detection of these individuals will enable personalized treatment to prevent and treat diabetes and its complications

DETAILED DESCRIPTION:
Breath samples will be collected in inert respiratory bag from diabetic and healthy volunteers, and analyzed using a chamber containing nano-chemical sensors. These samples together with blood samples will additionally be characterized using Gas Chromatography-Mass Spectroscopy "GC-MS".

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome
* Type 2 diabetes
* Healthy volunteers with 20<Body Mass Index<25

Exclusion Criteria:

* Smoking
* Chronic or acute lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Development of Diabetes or complication | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Karnieli, MD, Principal Investigator — Rambam Medicl Center, Technion
Locations (1):
- Rambam Medical Center - Inst. Endocrinology, Diabetes & Metabolism, Haifa, Israel